CLINICAL TRIAL: NCT00292656
Title: Importance of Hand Washing After Each NAET® Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nambudripad's Allergy Research Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: Hand washing After NAET; narfoundation study 119
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2006-04-04 (Estimated); Status verified 2006-02

CONDITIONS: Allergy
Keywords: Allergy
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Procedure: NAET

SUMMARY:
Background: It has been suspected in our clinic patients that when patients do not wash their hands after receiving NAET treatments, the effect of their treatments has been reduced or in some cases, the same treatment has to be repeated more times to be effective.

Location of the study: PNIB Research Center 6714 Beach Blvd. Buena Park, CA 90621

Purpose The purpose of the study was to determine the importance of hand-washing with plain water after each NAET® treatment. The study utilized an experimental design with random assignment to two groups, consisting of treatment/experimental, and treatment/control groups.

Objective: We sought to determine if there is any benefit to mandate hand-washing with plain water after each NAET® treatment.

DETAILED DESCRIPTION:
Selection of the Subjects:

The study was limited to the established patients in our clinic who came for NAET treatments on a Wednesday. Wednesday was chosen since it was a full working day and more patients will be treated on Wednesdays. First patient who arrived in the office was assigned into the experimental/treating group, then every odd number was selected as treating group. All even numbers were selected as placebo group..

Inclusion Criteria The primary inclusion criterion was that patients are getting treated for NAET on that day. All new patients were excluded. Only existing patients were chosen for this study. All the subjects included were required to sign a consent form, which allowed the researcher to designate them as subjects for the study.

Exclusion Criteria The exclusion criteria were: Serious illness, e.g., cancer, chronic obstructive pulmonary diseases, kidney diseases, heart diseases, pregnancy, mental diseases, and history of anaphylaxis.

Group Assignments:

38 females, and 22 males ages ranged between 12-60 years were randomly assigned to 2 groups:

1. Experimental group: 30 (22 females and 8 males) subjects were assigned to this group.
2. Control group: 30 (16 females and 14 males) subjects were assigned to this group.

Experimental Subjects:

They were advised to wash their hands with soap and water before beginning of NAET treatments. They were also asked to wash their hands with plain water (no soap) after completing NAET treatment before they left the office.

Control group:

They were advised not to wash their hands before or after the NAET treatment. They were allowed to go home soon after the treatment.

Evaluation Methods:

All subjects were treated for their appropriate scheduled allergens for that day. After the NAET, they waited for 20 minutes in the office. Then they were rechecked for the treated allergens. All of them had successfully completed their treatments. The experimental group was advised to wash their hands with plain water and they were advised to go home. The control group was advised to go home without washing their hands with water. They were asked to return on the following Wednesday for reexamination. A week after the treatment, they all returned for recheck and the resuls were recorded.

Duration of The Study The study duration was 7 days.

Results:

Experimental Group: 28 passed the treatment. 2 failed the treatment. Control Group: 5 passed the treatment. 25 failed the treatment. NAET Treatment was successful in 93.3% of the experimental group who utilized hand-washing after NAET treatment. NAET Treatment was successful 16.6% in the control group who did not wash their hands after NAET treatment.

Conclusion: The study concluded that hand-washing with plain water after each NAET treatment is essential for completing NAET treatments successfully.

Reprints Request from:

NAR Foundation 6714-32 Beach Blvd. Buena Park, CA 90621 narfoundation@yahoo.com

ELIGIBILITY:
Inclusion Criteria:

Allergy -

Exclusion Criteria:

None

-

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-12; Study Completion 2005-12

PRIMARY OUTCOMES:
We sought to determine if there is any benefit to mandate hand-washing with plain water after each NAET® treatment.

SECONDARY OUTCOMES:
Educational

CONTACTS AND LOCATIONS:
Overall Officials: Devi S. Nambudripad, DC,LAc.,PhD., Principal Investigator — NAR Foundation
Locations (1):
- 6714 Beach blvd., Buena Park, California, United States